CLINICAL TRIAL: NCT04292145
Title: Efficacy of an Application as a Relaxation Technique
Brief Title: Effectiveness of Relaxation Techniques
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sarah Corner (Other)
Responsible Party: Sponsor-Investigator, Sarah Corner, Principal Investigator, Southern Methodist University
Organization: Southern Methodist University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: H19-130-MEUA
Record Dates: First submitted 2020-02-07; First posted 2020-03-02 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Stress, Psychological
Keywords: breathe; breathing; relax; relaxation; respiration; stress
MeSH Terms: conditions — Stress, Psychological; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of the two groups as they enter the study.
Who Masked: Participant
Masking Description: Participants will not be aware of the purpose of the study, thus they will not know if they are in the experimental or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relaxation Application (Experimental): Participants will follow the relaxation application.
  Interventions: Behavioral: Relaxation Application
- Relaxation Only (Active Comparator): Participants will use any relaxation technique they normally use to relax.
  Interventions: Behavioral: Relaxation Only

INTERVENTIONS:
Behavioral: Relaxation Application — The use of an application for relaxation.
  Arms: Relaxation Application
Behavioral: Relaxation Only — The individual's personal method to relax.
  Arms: Relaxation Only

SUMMARY:
The study aims to assess the validity of a relaxation app. This will be accomplished by obtaining self-report measures about mood and respiratory symptoms. We hypothesize that self-report in the relaxation app condition will be different from that of the relaxation only condition.

ELIGIBILITY:
Inclusion Criteria:

* Student enrolled in SMU
* Speaks English

Exclusion Criteria:

* Must have an Apple Watch to use during time of participation in the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-04-22 (Actual); Primary Completion 2024-04-22 (Estimated); Study Completion 2024-12-22 (Estimated)

PRIMARY OUTCOMES:
Sensations Questionnaire | at study completion, up to 2 years
  Perceived bodily sensations. Scores range from 10-100, where higher scores indicate sensitivity to bodily sensations.
Positive and Negative Affect Schedule | at study completion, up to 2 years
  Immediate experience of mood. The measure consists of two scales, negative and positive items. Scores range from 10-50 for the positive scale, where higher scores indicate greater positive mood, and scores range from 10-50 for the negative scale, where higher scores indicate greater negative mood.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Y Kim, BA, Principal Investigator — Southern Methodist University
Locations (1):
- Southern Methodist University, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No